CLINICAL TRIAL: NCT03588299
Title: A Phase 1/2 Open-label Safety and Dose-finding Study of BAY2599023 (DTX201), an Adeno-associated Virus (AAV) hu37-mediated Gene Transfer of B-domain Deleted Human Factor VIII, in Adults With Severe Hemophilia A
Brief Title: Study to Test the Safety and How Well Patients With Severe Hemophilia A Respond to Treatment With BAY 2599023 (DTX 201), a Drug Therapy That Delivers a Healthy Version of the Defective Factor VIII Gene Into the Nucleus of Liver Cells Using an Altered, Non-infectious Virus (AAV) as a "Shuttle"
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Ultragenix pharmaceutical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19429; 2023-505827-29-00 (Other: CTIS(EU)); 2017-000806-39 (EudraCT Number)
Record Dates: First submitted 2018-07-06; First posted 2018-07-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A
Keywords: Severe hemophilia A (<1% FVIII activity); Factor VIII gene therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY2599023 / (DTX201) (Experimental): Adult patients with severe hemophilia A, who have been previously treated with FVIII products
  Interventions: Drug: BAY2599023 (DTX201)

INTERVENTIONS:
Drug: BAY2599023 (DTX201) — Single escalating doses with 4 dose steps; Single intravenous (IV) administration.

SUMMARY:
In this study researchers want to gather more information about safety and effectiveness of BAY 2599023 (DTX201), a drug therapy that delivers the human factor VIII gene into the human body by use of a viral vector to treat the disease. By replacing the defective gene with a healthy copy the human body may produce clotting factor on its own. Hemophilia A is a bleeding disorder in which the human body does not have enough clotting factor VIII, a protein that controls bleeding. Researcher want to find the optimal dose of BAY 2599023 (DTX201) so that the body may produce enough clotting factor on its own.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18 years or older.
* Confirmed diagnosis of hemophilia A as evidenced by their medical history with plasma FVIII activity levels < 1% of normal or at screening.
* Have >150 exposure days (EDs) to FVIII concentrates (recombinant or plasma-derived).

If on prophylaxis, are required to be willing to stop prophylactic treatment at specified time points throughout the study or If on-demand: should have had > 4 bleeding events in the last 52 weeks

- Agree to use reliable barrier contraception.

Exclusion Criteria:

* History of allergic reaction to any FVIII product.
* Clinically relevant findings in the physical examination considered critical by the treating physician, including obesity with BMI > 35 kg/m*2
* Current evidence of measurable inhibitor against factor VIII, prior history of inhibitors to FVIII protein or clinical history suggestive of inhibitor.
* Evidence of active hepatitis B or C.
* Currently on antiviral therapy for hepatitis B or C.
* Significant underlying liver disease.
* Serological evidence of HIV-1 or HIV-2 with CD4 counts ≤200/mm*3; HIV+ and stable participants with CD4 count >200/mm*3 and undetectable viral load are eligible to enroll.
* Detectable antibodies reactive with AAVhu37capsid.
* Participant with another bleeding disorder that is different from hemophilia A (e.g., von Willebrand disease, hemophilia B).
* Participated in a gene transfer trial within the last 52 weeks or in a clinical trial with an investigational product within the last 12 weeks.
* Known or suspected hypersensitivity or allergic reaction to trial product(s) or related FVIII products or any component of BAY2599023 (DTX201), or a contraindication to prednisolone

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2026-11-03 (Estimated); Study Completion 2026-11-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs), treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and AEs/SAEs of special interest | Up to 5 years.

SECONDARY OUTCOMES:
Expression pattern of FVIII activity. | Up to 5 years
  Determined using both a one-stage assay and chromogenic assay.
Proportion of patients in the respective dose step, that reached an expression of FVIII above 5% | At 6 months and 12 months following the IV administration of BAY2599023

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - Arkansas Children's Hospital - Hematology / Oncology, Little Rock, Arkansas
  - C.S. Mott Children's Hospital - Hematology / Oncology, Ann Arbor, Michigan
  - UW Health Carbone Cancer Center, Madison, Wisconsin
- SHATHD Spec. Hospi. for Active Treatm. of Haematol. Dis. EAD, Sofia, Bulgaria
- France (2):
  - APHP-Hopital Necker Enfants malades, Paris
  - CHU Rennes - Hopital Pontchaillou, Rennes
- Germany (2):
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Vivantes Klinikum im Friedrichshain, Berlin
- Netherlands (4):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medisch Centrum, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Manchester Royal Infirmary, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.